CLINICAL TRIAL: NCT02970578
Title: 3D-printed Module-assisted Minimally Invasive Lumbar Pedicle Screw Placement: a Retrospective, Self-controlled, Open-label Clinical Trial
Brief Title: 3D-printed Module-assisted Minimally Invasive Lumbar Pedicle Screw Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Principal Investigator, Haibin Lin, Chief Physician, The Affiliated Hospital of Putian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PutianU_001
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Thoracolumbar; Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3D printed module (Experimental): The patients underwent 3D printed module-assisted lumbar pedicle screw placement using the Quandrant system, aiming to restore the stability of the spine.
  Interventions: Procedure: 3D printed module

INTERVENTIONS:
Procedure: 3D printed module — The patients underwent 3D printed module-assisted lumbar pedicle screw placement using the Quandrant system, aiming to restore the stability of the spine.

SUMMARY:
To explore the accuracy of 3D printed module assisted minimally invasive lumbar pedicle screw placement using Quandrant system, and verify its feasibility of reducing error rate of screw placement and postoperative complications.

DETAILED DESCRIPTION:
History and current related studies Pedicle screw fixation has been widely used in spinal surgery, such as spinal fractures, lumbar spondylolisthesis, scoliosis, lumbar spinal stenosis. However, difficulties in pedicle screw placement are unavoidable because of anatomical variations in the spinal structure and spinal degeneration. Consequently, the precise localization for screw placement is essential. If not, errors in screw placement will result in reduced strength or even failure of the internal fixation, which may lead to a series of injuries, including nerve root injury, dural sac tear, vascular injury and even spinal cord injury. To conclude, it is urgent to improve the accuracy of screw placement and reduce complications of screw placement in the pedicle screw fixation.

With the rapid adoption of digital medicine and 3D printing technology in orthopedic practice, 3D techniques, based on preoperative high-resolution CT scan data, can theoretically restore the three-dimensional structure of the bone. That is to say, the investigators can present a detailed description of the complex anatomical structure of the bone, to accurately make a preoperative plan and an intraoperative simulation. Numerous evidences have been achieved with digital three-dimensional reconstruction and 3D techniques to assist the posterior pedicle screw fixation in the treatment of spine lesions.

Adverse events Postoperative adverse events were recorded and reported to the Affiliated Hospital of Putian Hospital within 24 hours.

Proper therapeutic measures could be performed if the following adverse events occurred, including incision infection, back muscle pain, dural sac tear, vascular injury, nerve root injury, spinal cord injury, screw falling off and loosening.

Data collection, management, analysis, and open access Baseline data were collected at the day when the participants were enrolled in the study. Other data were collected preoperatively, intraoperatively, postoperatively and during the follow-up. All data were input using Epidata and saved electronically.

All data regarding this clinical study were preserved by the Affiliated Hospital of Putian University, China.

All data were statistically analyzed by professional statisticians who were responsible for completing an outcome analysis report that was submitted to the project manager who was responsible for completing a research report. An independent data monitoring committee was responsible for data monitoring and management throughout the entire trial.

Statistical analysis All data were statistically analyzed by statisticians using SPSS 19.0 software (IBM Corporation, Armonk, NY, USA) in accordance with the intention-to-treat principle.

Normally distributed measurement data were expressed as means, standard deviations, minimums, and maximums; non-normally distributed data were expressed as lower quartiles, medians, and upper quartiles.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar degenerative diseases as diagnosed by the criteria for diagnosis of lumbar degenerative diseases
* Indications for internal fixation in the degenerative lumbar spine
* Lumbar single segment or multi-segment lesions
* Average age 63 years
* Provision of the informed consent

Exclusion Criteria:

* Lumbar spine tumors, lumbar tuberculosis, trauma fractures or joint disorders
* Lumbar infection or acute inflammation in the other parts of the body
* Unable to undergo lumbar surgery due to surgical contraindications (coagulation disorders) and poor cardiopulmonary function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Accurate rate of screw placement | during the operation
  To assess whether the screw placement by 3D printed module navigation achieves the desired results. The higher value indicates the higher accuracy.

SECONDARY OUTCOMES:
Lumbar CT imaging | Baseline and month 6, month 24 after surgery
  To observe the conditions of lumbar fixation.
Time of operation | during the operation
  To evaluate the speed of surgery. The shorter operation time indicates that this method is easier to operate.
Amount of intraoperative bleeding | during the operation
  To evaluate the conditions of intraoperative blood loss. Less blood loss indicates the higher improvement in the surgical quality by this method being studied.

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Lin, bachelor, Principal Investigator — The Affiliated Hospital of Putian University

IPD SHARING:
Plan to Share IPD: Undecided